CLINICAL TRIAL: NCT03039296
Title: EuroPainClinics® Study IV (Prospective Observational Study)
Acronym: EPCSIV
Status: Terminated | Type: Observational
Why Stopped: The low number of participants was enrolled in to the clinical trial
Sponsor: Europainclinics z.ú. (Other)
Responsible Party: Sponsor
Other Study IDs: 5N/2016
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Low Back Pain; Facet Joint Pain
Keywords: Low back pain; Facet joints; Endoscopic rhizotomy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- One side endoscopic rhizotomy: Endoscopic rhizotomy will be provided only on one back side according pain
  Interventions: Procedure: Endoscopic rhizotomy
- Both sides endoscopic rhizotomy: Endoscopic rhizotomy will be provided on both back sides according pain
  Interventions: Procedure: Endoscopic rhizotomy

INTERVENTIONS:
Procedure: Endoscopic rhizotomy — Endoscopic rhizotomy (facet joint denervation) is carried out through the insertion of an endoscope to the medial spinal nerve area with the help of mobile C-arm x-ray guidance. The tissue surrounding the medial nerves is endoscopically visualized and dissected with a sterile grasper to expose the nerve structure. Finally, a radiofrequency probe is used to ablate the problematic medial branch nerve under direct endoscopic control. The procedure is concluded with the removal of the endoscope and the small incision is closed with 1-2 skin sutures.

SUMMARY:
In this prospective observational trial the effect of the Endoscopic rhizotomy microinvasive therapy should be examined in (approximately 150) adult patients with low back pain positive for facet joint pain component.

DETAILED DESCRIPTION:
Facet joint pain encompasses a significant portion of possible sources of pain in patients with vertebrogenic algic syndrome. A typical symptom is intermittent radiation of pain in the back and legs. The cause of this pain is irritation of the medial branch of the dorsal nerve root, which innervates a facet joint. Confirmation of the source of pain involves using a local anaesthetic to block the medial branches of several vertebral areas. If, through this test, the facet joints are determined to be the source of pain the patient's condition is indicated for radiofrequency ablation of the nerve branches.

EuroPainClinics® Study IV (EPCS IV) is a prospective observational comparative study that will use pain scales to analyse changes in the neurological status of nerves of patients who undergo the minimally invasive procedure: radiofrequency nerve ablation and cryoablation of the lumber facet joints.

The study aims to investigate documented clinical results of the neurological conditions of patients, to compare pain scales and the use of analgesics over a number of time periods: prior to the procedure, 6 weeks post-procedure, as well as 6 and 12 months post-procedure. The data will be subsequently statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo Endoscopic rhizotomy therapy

Exclusion Criteria:

* No

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to investigate documented clinical results of the neurological conditions of patients, to compare pain scales and the use of analgesics over a number of time periods: prior to the procedure, 6 weeks post-procedure, as well as 6 and 12 months post-procedure. The data will be subsequently statistically analysed.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by the Visual analogue scale | 4 years
  All acquired information will be noted in to the special anonymous protocol

SECONDARY OUTCOMES:
Pain localization as assessed by note of radiating dermatome as neurologic examination | 4 years
  All acquired information will be noted in to the special anonymous protocol
Pain progress as assessed by global pain scale | 4 years
  All acquired information will be noted in to the special anonymous protocol
Changes in analgesics drugs consumption as assessed by equianalgesic dose ratios for opioids | 4 years
  All acquired information will be noted in to the special anonymous protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ladislav Kočan, MD PhD, Study Director — europainclinicsstudy@gmail.com
Locations (1):
- Europainclinics, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided